CLINICAL TRIAL: NCT04789070
Title: A Double-Blind Randomised Controlled Trial (dbRCT) Phase III Trial Investigating the Effect of Sirolimus on Disease Progression in Patients With Inclusion Body Myositis (IBM) as Measured by the IBM Functional Rating Scale (IBM-FRS)
Brief Title: Phase III Trial of Sirolimus in IBM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: The Perron Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Optimism in IBM
Record Dates: First submitted 2021-02-15; First posted 2021-03-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Active Comparator): 2mg capsules once daily
  Interventions: Drug: Sirolimus
- Placebo (Placebo Comparator): 2mg capsules once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Sirolimus is a currently licensed drug primarily used for immunosuppression post-kidney transplantation to prevent organ rejection. Sirolimus was initially considered as a treatment in IBM for its immunosuppressive action and beneficial effects in an experimental myositis mouse model.(11) Transfer of effector T cells from affected to healthy animals resulted in myositis, but the presence of Treg cells were protective against development of myositis. As Sirolimus, which acts to deplete effector T cells but preserving the Treg cells, was effective in this mouse model of myositis, it was therefore postulated that it may also be effective in IBM, not only for its effects on effector T cells and Treg cells, but also for its additional effects on protein degradation.
  Other Names: Rapamune
  Arms: Sirolimus
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The hypothesis is that Sirolimus, (Rapamycin (R)) which is currently used in organ transplantation and works by blocking the activity of T effector cells but preserving T regulatory cells, as well as by inducing autophagy (protein degradation), will be effective in IBM to slow or stabilize disease progression, helping to maintain patient function and independence. This phase III trial will confirm pilot data showing statistically significant clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults able to read and understand the Participant Information Sheet, and who freely provide written Informed Consent for the study;
2. Males or females aged 45 years or older;
3. Diagnosis of IBM according to the criteria proposed by the ENMC criteria 2011;
4. Able to walk a minimum distance of 200m within 6 minutes (walking aids, including frames, may be used);
5. Evidence of disease progression over the previous 12 months, as determined by a neuromuscular specialist through patient history, physical examination, MMT, IBM-FRS or other metrics.

Exclusion Criteria:

1. Inability to complete a 6MWT with a minimum distance of 200m achieved;
2. Inability to complete a mTUG or any other study procedure, including inability to swallow study drug, or clinical suspicion that the participant will become unable to swallow the study drug during the study period;
3. Unwillingness or inability to comply with study interventions or study schedule;
4. Hypersensitivity to Sirolimus, Everolimus or any compound of the oral solution;
5. Any prior exposure to Sirolimus or Everolimus within the last 6 months;
6. Presence of any other clinically significant disease that might interfere with patients ability to comply with study procedures, or places the patient at greater risk for SAEs;
7. Clinical suspicion of moderate or severe respiratory insufficiency based on history, clinical examination or respiratory function tests with an FVC < 50% of predicted; Nocturnal NIV is allowed for sleep-disordered breathing;
8. Severe chronic kidney disease or renal insufficiency with proteinuria (e.g Estimated Glomerular Filtration Rate < 30 ml/min and/or proteinuria as defined by spot urine protein/creatinine ratio > 100mg/mmol;
9. Chronic liver disease (cirrhosis and/or ALT/AST > 3 times the upper limit of normal (ULN)) , excluding cases in which raised ALT/AST are deemed to be due to underlying muscle disease. Patients can be re-screened within the window if a one-off measurement is elevated due to an acute injury such as a viral infection;
10. History of cancer (Except localised skin cancers including BCC/SCC) during the past 5 years;
11. Systemic autoimmune or rheumatological disease not in remission and/or necessitating specific treatment during the last 12 months. This includes significant organ-specific autoimmune disorder (e.g Grave's disease) not in remission and/or necessitating specific treatment during the past 12 months;
12. Any unhealed wounds or active infections at the time of screening;
13. If patient has received a live vaccine within the last 12 weeks;
14. Participants must be HIV negative, and Hepatitis C Virus Ribonucleic Acid (HCVRNA) Polymerase Chain Reaction (PCR) negative, and Hep B surface antigen negative and Hep B core antibody negative;
15. One or more the following blood test results at screening:

    1. Total cholesterol > 8 mmol/l (304mg/dl)
    2. Triglycerides > 5 mmol/l (>194 mg/dl)
    3. Haemoglobin < 110 g/L (11g/dl)
    4. Platelet count < 100 x 109/L
    5. Neutrophils < 1.5 x 109/L
    6. Lymphocytes < 1.0 x 109/L
16. Presence at screening of any medically significant cardiac, neurological, pulmonary, gastrointestinal, musculoskeletal or psychiatric illness (including uncontrolled anxiety and/or depression) that in the Investigator's opinion might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety or IBM-FRS;
17. Has taken any investigational study drug within 30 days or five half-lives of the prior agent (whichever is longer) prior to the Baseline visit;
18. Patient taking any other immunosuppressive or immunomodulatory medication (including but not limited to prior high dose prednisolone (>10mg/day) in the last 4 weeks, Intravenous Immunoglobulin (IVIG) within the last 3 months, methotrexate, mycophenolate, Sirolimus, Everolimus, calcineurin inhibitors, (cyclosporine or tacrolimus) or azathioprine within the last 6 months, and rituximab, alemtuzumab or other biologics within the last 12 months);
19. Other medications or products that may affect the metabolism of Sirolimus (See concomitant medications in Section 27) such as the following at time of screening:

    1. Strong inhibitors of CYP3A4 and/or P-gp (eg ketoconazole, voriconazole, itraconazole, telithromycin, erythromycin or clarithromycin)
    2. Strong inducers of CYP3A4 and/or P-gp (eg rifampicin, rifabutin, Phenytoin, Phenobarbitol, St John's Wort);
20. Use of any investigational drug other than study medication;
21. Pregnancy or planning a pregnancy:

    1. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test prior to randomisation, and must have a negative urine pregnancy test within 24 hours prior to the start of study drug. WOCBP must agree to use 'highly effective' contraception (MHRA guidelines, 2014) for the duration of the study and for 12 weeks post-treatment completion.
    2. Men who are sexually active with a WOCBP must agree to use barrier contraception (condom) for the duration of treatment with study drug and for 30 days post-treatment completion.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in IBM Functional Rating Scale (IBM-FRS) from Baseline to Week 84 | Baseline, Week 84
  The IBM-FRS is a concise and quick (~10 minute), clinician-administered ordinal rating scale used to determine participants' assessment of their capability and independence. It includes 10 measures (swallowing, handwriting, cutting food and handling utensils, fine motor tasks, dressing, hygiene, turning in bed and adjusting covers, changing position from sitting to standing, walking, and climbing stairs), graded on a Likert scale from 0 (being unable to perform) to 4 (normal). The sum of the 10 items gives a value between 0 and 40, with a higher score representing less functional limitation.

SECONDARY OUTCOMES:
Change in 6 Minute Walk Test (6MWT) from Baseline to Week 84 | Baseline, Week 84
  The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance in patients with cardiopulmonary disease. It is now a commonly used and validated test to estimate the functional walking capacity in patients with a range of chronic diseases including IBM.
Change in Modified Timed Up and Go (mTUG) from Baseline to Week 84 | Baseline, Week 84
  The Timed Up and Go (mTUG) was initially developed as a tool to determine falls risk, mobility, balance and walking ability in an elderly population. It has since been adopted as an outcome measure in a broader clinical setting including myositis.
Change in Manual Muscle Testing (MMT) from Baseline to Week 84 | Baseline, Week 84
  Manual Muscle Testing (MMT) is a relatively simple method of assessing a patient's strength in a muscle or group of muscles. There is however a degree of subjectivity when assigning a score. MMT will be used to assess change in strength throughout the study period. This method is routinely performed in a clinical setting and has been shown to be reliable. This tool assesses muscle strength using a 0 - 10 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Dimachkie, Principal Investigator — University of Kansas Medical Center
Locations (10):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
- Australia (7):
  - Concord Repatriation Hospital, Sydney, New South Wales
  - Royal Northshore Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria
  - Perron Institute, Perth, Washington
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badrising UA, Henderson R, Reddel S, Corbett A, Liang C, Reardon K, Ghaoui R, Bulsara M, Brady S, Brusch A, Chan D, Coudert JD, Fairchild T, Jain G, Kiernan MC, Leonard D, Lloyd T, Schmidt J, McDermott MP, Sanders L, Lowe C, van der Kooi AJ, Weihl C, Mohassel P, Simpson M, Carroll A, Cooper I, Beer K, Hiscock K, Walters S, Panicker A, Doverty A, Heim A, van Heur-Neuman M, Benveniste O, Dimachkie MM, Needham M. Optimism in inclusion body myositis: a double-blind randomised controlled phase III trial investigating the effect of sirolimus on disease progression in patients with IBM as measured by the IBM Functional Rating Scale. Clin Exp Rheumatol. 2025 Feb;43(2):316-325. doi: 10.55563/clinexprheumatol/zvffa0. Epub 2025 Feb 26. PMID 40018746